CLINICAL TRIAL: NCT05338203
Title: Comparison of Breast Milk Contents in Tandem Breastfeeding and Non-Tandem Breastfeeding Mother
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sidika Pelit Aksu, Research asistant (RN), Gazi University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 10840098
Record Dates: First submitted 2022-03-30; First posted 2022-04-21 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Tandem Breastfeeding
Keywords: mother milk; Breastfeeding; tandem
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (tandem breastfeeding) (Experimental): mother mılk wıll collected from these mother and they wıll be analyzed
  Interventions: Other: tandem breastfeedıng
- control group ( non-tandem breastfeeding) (No Intervention): mother mılk wıll collected from these mother and they wıll be analyzed

INTERVENTIONS:
Other: tandem breastfeedıng — mother mılk wıll collected from mothers and they wıll be analyzed in laboratuar.
  Arms: experimental group (tandem breastfeeding)

SUMMARY:
Breastfeeding is the gold standard for feeding newborns and infants. Tandem breastfeeding is defined as breastfeeding during pregnancy or simultaneous breastfeeding of two non-twins. The aim of this study; The aim of this study is to compare breast milk contents of mothers who breastfeed in tandem and mothers who do not breastfeed in tandem. The study was planned as an experimental study with a single center control group. The place where the research will be conducted is the Lactation/Relactation outpatient clinic and gynecology and obstetrics polyclinic of Çamlıca Medipol University Hospital and Halil Şıvgın Çubuk State Hospital. and tandem non-breastfeeding mothers. Power analysis was performed to determine the number of samples. For this purpose, the study results of Rosenberg et al. (2021) (Experiment: 8.1±0.2 Control:6.2±1.5) were used as reference. According to the power analysis made by calculating the effect size, the sample size calculated with α= 0.01 error level and 99% power; 18 women in the experimental group and 18 women in the control group, a total of at least 36 women. The analysis was made in G*Power version 3.1.9.4. All mothers will be informed about the study, and mothers who accept the study will have to fill out the "Conformity to Criteria Form" created by the researchers. Written informed consent will be obtained from mothers who meet the research criteria. After completing the introductory information form, milk will be collected from all mothers. Milk collection will be done by one of the researchers. Milking will always be collected from all mothers between 08:00 and 16:00, provided that at least 40 minutes have passed after the last milking. Manual milking will be done for 10 minutes.

DETAILED DESCRIPTION:
There are studies on the concentration of macronutrients in breast milk in the literature A few studies have examined macronutrients in breast milk in mothers who breastfeed in tandem. Sinkiewicz-Darol et al. (2021) in his study; Macronutrients in breast milk in mothers who breastfeed in tandem have been studied. Breast milk during tandem breastfeeding had higher fat content, energy value, and total protein concentration than milk after weaning the older child. The carbohydrate content remained constant. In the study of Rosenberg et al., (2021), the concentration of macronutrients in breast milk was investigated in tandem breastfeeding and non-tandem breastfeeding mothers. As a result, it was determined that breast milk produced during pregnancy has different macronutrient content than breast milk produced after birth. It was determined that colostrum and mature milk of mothers who breastfed in tandem were similar to the milk of mothers who did not breastfeed in tandem, except for the carbohydrate content. Breastfeeding and tandem breastfeeding during pregnancy have not been extensively studied. For this reason, our study will determine the effect of tandem breastfeeding on the macronutrient content of breast milk and will provide evidence for tandem breastfeeding, which is traditionally practiced by many women.

1.2 Purpose of Research The aim of this study; The aim of this study is to compare the breast milk contents of tandem breastfeeding and non-tandem breastfeeding mothers.

2. METHODS and MATERIALS 2.1. Type of Research The research was planned as an experimental study with a single center control group.

2.2. Place of Research The place where the research will be carried out is the Lactation/Relactation polyclinic and gynecology and obstetrics polyclinic of Çamlıca Medipol University Hospital and Halil Şıvgın Çubuk State Hospital.

2.3. Sample of the Research The population of the study will be tandem breastfeeding and non-tandem breastfeeding mothers who applied to the Lactation/Relactation outpatient clinic of Çamlıca Medipol University Hospital and Halil Şıvgın Çubuk State Hospital, and the obstetrics and gynecology outpatient clinics. Power analysis was performed to determine the number of samples. For this purpose, the study results of Rosenberg et al. (2021) (Experiment: 8.1±0.2 Control:6.2±1.5) were used as reference. According to the power analysis made by calculating the effect size, the sample size calculated with α= 0.01 error level and 99% power; 18 women in the experimental group and 18 women in the control group, a total of at least 36 women. The analysis was performed in G*Power version 3.1.9.4.

2.3.3. Example Selection Criteria All women who meet the following criteria will be invited to participate in the study.

Experiment:

* If pregnant, being in the second trimester of pregnancy; have given birth, postpartum 16th day or more
* If pregnant, not having a risky pregnancy
* If she is pregnant, there is a report from the obstetrician she is followed that there is no harm in breastfeeding
* The older child being breastfed is under the age of 2
* Absence of literacy problems, mental disabilities and communication problems
* Absence of chronic disease
* No communicable disease
* Not using a drug continuously
* Not using any medication in the last 24 hours
* Willingness to participate in the study

Control:

* Postpartum 16th day and above
* No risky pregnancy in her last pregnancy
* Being multiparous
* Absence of literacy problems, mental disabilities and communication problems
* Absence of chronic disease
* No communicable disease
* Not using a drug continuously
* Not using any medication in the last 24 hours
* Willingness to participate in the study During the research process, mothers will be excluded from the sample in case the mothers want to leave the study, the sample milk is spoiled or there are losses during the analysis.

2.3.4. Randomization Randomization will not be possible in the study. 2.4. Data Collection All mothers will be informed about the study, and mothers who accept the study will have to fill out the "Conformity to Criteria Form" created by the researchers. Written informed consent will be obtained from mothers who meet the research criteria. After completing the introductory information form, milk will be collected from all mothers.

Collection of breast milk Milk collection will be done by one of the researchers. Milking will always be collected from all mothers between 08:00 and 16:00, provided that at least 40 minutes have passed after the last milking. Manual milking will be done for 10 minutes.

Collected breast milk samples will be frozen at -180C within two hours. It will be allowed to dissolve by keeping it at +40C 48 hours before the analysis. Breast milk samples, which are heated up to 400C in a water bath, will be homogenized by Miris Ultrasonic Homogenizer for 5 seconds just before analysis. Breast milk samples will be analyzed with Miris®️ HMA, and protein, fat, carbohydrate and energy values will be determined. Miris®️ HMA (Uppsala, Sweden) is certified by the International Standards Organization (ISO) 9622: 1999. The device, which has different filters for special milk components, uses four different wavebands for fat, protein and lactose determination. Miris®️ HMA device consists of a cuvette and auxiliary equipment. The so-called cuvette is a mid-infrared measuring cell with an inlet and an outlet. Breast milk is injected through the vestibule, passing through two CaF2 windows divided by a spacer (50 μm). On one side of the windows is a source of infrared radiation (emitter) and on the other side there is a four-channel detector that receives the radiation transmitted through the liquid. The filters in the detector are chosen to absorb mid-infrared radiation associated with fat, protein and carbohydrate. The fourth filter acts as a reference filter. Radiation from the infrared source passes through the Transparent cuvette with the liquid sample, assessing the amounts of radiation absorbed by specific functional groups of fat, protein and carbohydrate, respectively. The quantitative determination of fat, protein and carbohydrate absorbed in direct proportion to the concentration is made according to Beer's law. Each macronutrient composition is calculated by Miris®️ HMA in g per 100 ml. Fat molecules are determined by ester bonds to the carbonyl groups of glycerides, and protein molecules are determined by the infrared method with the second amide group of peptide bonds. The lactose content is analyzed by lactose and hydroxyl groups of mono/oligosaccharides, and the total energy is determined by calculating the measurement results. The pH measurement will be measured with the MW102, Milwaukee® instrument.

2.4.1. Data Collection Tools 'Conformity to Criteria Form' (Appendix-1), Introductory Information Form (Appendix-2) and 'Breast Milk Biochemical Analysis Form' (Appendix-3) will be used in collecting research data.

2.4.1.1. Conformity to Criteria Form (Annex-1) This form includes a checklist of inclusion criteria. 2.4.1.2. Introductory Information Form (Appendix -2) This form, which was developed by the researcher using the literature, has 5, which determines the socio-demographic characteristics of mothers (age, education level, income level, occupation), 6 that determines their obstetric characteristics (number of pregnancy, gestational week, birth), and 1 is about the baby and breastfeeding, a total of 12 forms. consists of questions.

2.4.1.3. Breast Milk Biochemical Analysis Form (Appendix-3) Developed by researchers. In the evaluation of breast milk content, Ph, fat, carbohydrate, protein and energy values, which are possible to change with the milking method, will be written on the form according to the results of the analysis.

2.5. Evaluation of Data The data obtained in the research will be evaluated with the SPSS (Statistical Package of Social Sciences) 22.0 package program. The homogeneity of the variances in both groups will be checked with the Levene test, and the normality with the Shaphiro Wilk test. If the variances are homogeneous and normally distributed, T-test will be used for independent groups from parametric tests, and if the variances are not homogeneous and do not show normal distribution, the Mann Whitney-U test will be used. 0.05 will be used as the level of significance and it will be stated that there is a significant relationship in case of p<0.05, and that there is no significant relationship in the case of p>0.05. In order to determine the effect of mediator variables on breast milk, mediator and moderator variable analyzes will be performed.

2.6. Ethical Aspect of Research The application will be started after the necessary permissions from the institution where the research will be conducted, the ethics committee and written consent from the mothers are obtained. Mothers can opt out of the study whenever they want. No payment will be made to mothers for participating in the study.

ELIGIBILITY:
Inclusion Criteria of Experiment Group:

* If pregnant, being in the second trimester of pregnancy; have given birth, postpartum 16th day or more
* If pregnant, not having a risky pregnancy
* If she is pregnant, there is a report from the obstetrician she is followed that there is no harm in breastfeeding
* The older child being breastfed is under the age of 2
* Absence of literacy problems, mental disabilities and communication problems
* Absence of chronic disease
* No communicable disease
* Not using a drug continuously
* Not using any medication in the last 24 hours
* Willingness to participate in the study

Inclusion Criteria of Control Group:

* Postpartum 16th day and above
* No risky pregnancy in her last pregnancy
* Being multiparous
* Absence of literacy problems, mental disabilities and communication problems
* Absence of chronic disease
* No communicable disease
* Not using a drug continuously
* Not using any medication in the last 24 hours
* Willingness to participate in the study

Exclusion criteria. During the research process, mothers will be excluded from the sample in case the mothers want to leave the study, the sample milk is spoiled or there are losses during the analysis.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-04-15 (Estimated); Primary Completion 2022-05-15 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
change in protein levels | 15 days
  ıt wıll be analyzed from mılk

SECONDARY OUTCOMES:
change in ph levels | 15 days
  ıt wıll be analyzed from mılk
change in carbonhidrad levels | 15 days
  ıt wıll be analyzed from mılk
change in energy levels | 15 days
  ıt wıll be analyzed from mılk
change in fat levels | 15 days
  ıt wıll be analyzed from mılk

CONTACTS AND LOCATIONS:
Overall Officials: Sıdıka PELİT AKSU, PhD, Principal Investigator — Gazi University
Locations (1):
- Sıdıka PELİT AKSU, Ankara, Turkey/Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No